CLINICAL TRIAL: NCT06330116
Title: A Comparison of Three Different Forms of Oral Myofunctional Training (OMT) as Methods for Reducing Snoring and Mild to Moderate Sleep Apnea
Brief Title: Different Forms of OMT as Methods for Reducing Snoring and Mild to Moderate Sleep Apnea
Acronym: SNORT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västerbotten (Other Government)
Collaborators: Interreg (Other); Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-05348-01
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Sleep Apnea, Obstructive; Snoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Intervention Model Description: 141 consecutive adult subjects, 71 men and 70 women, referred to hospital, due to symptoms of snoring and mild to moderate sleep apnea will be randomized, included, and examined at three different sights, Umeå(Sweden), Lund(Sweden) and Köge(Denmark) One hundred-five of them, 35 in each treatment group, will receive one of the 3 different forms of training and the final 36 persons serving as controls, age/AHI matched (18 in Köge resp Umeå). Patients in Umeå will be randomized to either training with IQoro or serving as controls. Patients in Köge will be randomized to either training with Exciteosa group training, or controls.
Who Masked: Outcomes Assessor
Masking Description: The study will use a prospective randomized open-blinded endpoint (PROBE) design with baseline measurements, intervention phase and follow-up measurements, and controls without intervention. The results are then analyzed and blinded to the evaluators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Oral screen (Active Comparator): Strength training of the oral and pharyngeal muscles is performed with an oral screen (OS)(IQoro). The OS is a device that has an effect both on the brain plasticity and a strengthening effect of oral and pharyngeal muscles. (9) The OS is placed pre-dentally behind closed lips. The patient pulls the OS forward in a horizontal direction with strong pressure for 5 to 10 seconds while firmly resisting the pressure with tightened lips. The exercise is repeated three times, with 3 seconds of rest between repetitions, and is performed 3 times per day. Training for 3 months.
  Interventions: Device: IQoro
- Neuromuscular electrical training (NMES) (Active Comparator): Strength training of the oral and pharyngeal muscles is performed by an oral device used for 20 minutes every day (eXciteosa). The device gives electrical pulses to the surrounding tissue, mainly the tongue. Training for 3 months.
  Interventions: Device: eXciteosa
- Group training with an occupational therapist (Active Comparator): Strength training of the oral and pharyngeal muscles is performed in group, led by an occupational therapist. Training for 3 months.
  Interventions: Behavioral: Grouptraining

INTERVENTIONS:
Device: IQoro — Please refer to arm/group description for information
  Arms: Oral screen
Device: eXciteosa — Please refer to arm/group description for information
  Arms: Neuromuscular electrical training (NMES)
Behavioral: Grouptraining — Please refer to arm/group description for information
  Arms: Group training with an occupational therapist

SUMMARY:
Objective the present project aims to assess the impact of 1) oral screen training, group training, and the use of neuromuscular electrical training (NMES) as orofacial myofunctional therapy (OMT) methods for reducing the apnea-hypopnea index (AHI) among adults with mild to moderate sleep apnea and 2) if these different training methods can reduce snoring and affect the level of sleepiness and quality of life. Study design The study will use a prospective randomized open-blinded endpoint (PROBE) design with baseline measurements, intervention phase, and follow-up measurements.

Methods 141 consecutive adult subjects, 71 men and 70 women referred to hospital, due to symptoms of snoring and mild to moderate sleep apnea will be randomized, included, and examined at three different sites, Umeå(Sweden), Lund(Sweden) and Köge(Denmark) One hundred-five of them, 35 in each treatment group, will receive one of the three different forms of training and the final 36 persons serving as controls, age/AHI matched (18 in Köge resp Umeå). Participants in Umeå will be randomized to either training with IQoro® or serving as controls. Participants in Köge will be randomized to either training with Exciteosa®, group training, or controls.

The primary outcome is a change in AHI before and after three months of training with the different methods according to overnight ambulatory sleep apnea recordings.

The secondary outcomes are change in snoring frequency, sound level dB (A) according to a questionnaire, the Basic Nordic Sleep Questionnaire (BNSQ), daytime sleepiness using the Epworth Sleepiness Scale (ESS), change in quality of life using the short form -36 (SF-36) and muscle strength in tongue before and after treatment.

DETAILED DESCRIPTION:
Introduction/Background

Snoring and obstructive sleep apnea (OSA) are common among the adult population; a mean of 22% and 17% of the women are affected. Obstructive sleep apnea is related to several negative health effects, such as sleepiness, hypertension, cardiovascular disease, and cognitive impairment. Continuous positive airway pressure (CPAP), oral appliances (OA), as well as oropharyngeal surgery in selected cases are available as a treatment for OSA. The same methods can be used for reducing snoring, but the cost for the devices is high, and the compliance tends to be low, although snoring affects the individual as well as the bed partner. Snoring produces vibrations in the upper airway, and over time, it can affect both the motor and sensory function of the tissue in the upper airway. The deterioration process is unknown, but previously published data shows a correlation between the level of snoring/OSA and altered sensory and motor function. This is probably due to the adverse effects of the vibrations and stretching of the nerves and muscles in the airway during snoring and apneas. Our and other research groups have presented similar results and hypothesize that the deterioration may explain why the airway slowly tends to collapse more frequently. This may also explain why more than half of the habitual snorers show deviant swallowing function and thereby have a higher risk of aspiration. It is unknown if this degenerative process of the upper airway is possible to slow down, stop or perhaps even be reversed and thereby improve the sensory and motor function by treatment that decrease or determine snoring and OSA. However, recent data give promising indications that myofunctional training of the upper airway can decrease levels and intensity of snoring and reduce the apnea-hypopnea index (AHI).

Oral screen training can affect brain plasticity and have a strengthening effect on oral and pharyngeal muscles. Oral screen training is used to improve oral and pharyngeal muscle function and has been reported to improve swallowing function in patients suffering from dysphagia including aspiration after stroke. Further, it has been reported to be efficient for the treatment of dysphagia caused by other conditions.

Daily neuromuscular electrical training (NMES) by an oral device eXciteosa® has shown promising results in patients with primary snoring and mild sleep apnea, reducing objective and subjective snoring. Orofacial training guided by an occupational therapist (group training) has also shown positive results in adhering to the training program and affecting the AHI, reducing it in persons aged 60 and younger.

The aim of the present study is, therefore, to assess 1) the impact of three different training methods to reduce AHI among adults with mild to moderate sleep apnea and 2) if the oral screen training can lower the level and intensity of snoring, change levels of sleepiness, quality of life and strength of the tongue muscle.

Material and methods

Subjects and procedure In total 141 consecutive adult subjects, 71 men and 70 women, referred to Umeå University Hospital and Köge University Hospital, due to symptoms of snoring and/or mild to moderate sleep apnea, will be included. The subjects included in Umea will get three months of intervention with oral screen training or serve as controls. The subjects included in Köge will get either a three-month intervention with orofacial group training led by an occupational therapist, three months intervention with a daytime mouth device for muscular training, eXciteosa® or serve as controls. At baseline, all subjects will undergo two overnight ambulatory sleep apnea recordings and answer questionnaires regarding snoring, daytime sleepiness, and quality of life. The demography, including sex, age, and BMI, will be recorded. Tounge strength will be measured.

In Umeå, the participants will be randomly assigned to either an initial three-month intervention with oral screen training or a three-month intervention delay, serving as controls. In Köge, the participants will be randomly assigned to either a three-month intervention with eXciteosa®, group training with an occupational therapist, or serve as controls. After three months, all the above questions and parameters will be registered again.

Inclusion criteria are men and women with AHI 10 - 29 seeking for problems with snoring and obstructive sleep apnea, age 18 to 75.

Exclusion criteria are subjects with previous soft palate surgery, 9 < AHI > 29, smokers, New York Heart Association Functional Classification, NYHA ≥ 3. BMI >34,9.

Main outcome measurements The primary outcome is the change in the apnea-hypopnea index (AHI) before and after three months of training with one of the modalities.

Secondary outcome measurements The secondary outcomes are a change in snoring frequency and sound level dB (A) and a a questionnaire concerning snoring, the Basic Nordic Sleep Questionnaire (BNSQ).

Daytime sleepiness was assessed using the Epworth Sleepiness Scale (ESS) change in quality of life using the short form -36 (SF-36) and change in muscle strength before and after treatment.

Oral screen (Only in Sweden) Strength training of the oral and pharyngeal muscles is performed with an oral screen (OS)(IQoro®). The OS is a device that has an effect both on the brain plasticity and a strengthening effect of oral and pharyngeal muscles. The OS is placed pre-dentally behind closed lips. The participant pulls the OS forward in a horizontal direction with strong pressure for 5 to 10 seconds while firmly resisting the pressure with tightened lips. The exercise is repeated three times, with 3 seconds of rest between repetitions, and is performed 3 times per day.

Neuromuscular electrical training (NMES) (Only in Denmark) Strength training of the oral and pharyngeal muscles is performed by an oral device used for twenty minutes every day (eXciteosa®). The device gives electrical pulses to the surrounding tissue, mainly the tongue.

Group training with an occupational therapist (Only in Denmark) Strength training of the oral and pharyngeal muscles is performed in a group led by an occupational therapist.

Sleep apnea recordings The investigators will use two types of recording devices, Nox-T3® (Nox-T3®, Nox Medical Inc.

Reykjavik, Iceland) and SleepImage® System (MyCardio LLC, Denver, CO, USA) In the overnight home sleep studies, recordings will be scored manually (Nox-T3®), and the scorer is blinded to the treatment (blinded endpoint). All recordings will be done over two nights, at baseline and follow-up to minimize the effect of night-to-night variability.

The duration of sleep will be estimated from the recordings. An apnea is defined as a drop in the peak thermal sensor excursion of > 90 of the baseline lasting at least 10 seconds, while a hypopnea is defined as a 50% reduction in airflow compared with baseline, combined with an oxygen desaturation of > 3%.

Obstructive sleep apnea is defined as a mean of five or more obstructive apneas and hypopneas per hour of sleep. Mild sleep apnea is considered when the apnea-hypopnea index is 5 to < 15, moderate sleep apnea when the apnea-hypopnea index is 15 to < 30, and severe sleep apnea when the apnea-hypopnea index is > 30.

The snoring frequency and sound level dB (A) will be measured with a microphone within the recording device (Nox-T3®) and a questionnaire regarding the level and frequencies of the snoring (BNSQ).

Additionally, the investigators will also use a new device called Sleepimage®. The device measures plethysmography trace, heart (pulse) rate, heart (pulse) rate variability, respiration, blood oxygenation (SpO2), and actigraphy. The device is a ring worn on any finger on the left hand and collects sleep data during the night. The result is then translated into a report giving data about sleep quality, any sleep pathology, and sleep duration. The device has FDA approval At present, there is no "golden standard" for measuring snoring. However, the methods and devices have improved, and a recent comparison of different tools for measuring snoring suggested the use of the T3 advice for the recordings.

Measuring strength:

Tounge strength is measured with the Iowa Oral Performance Instrument, IOPI®.

Questionnaires:

The Basic Nordic Sleep Questionnaire (BNSQ) BNSQ was developed in Nordic countries to develop a standardized questionnaire. The task force developing it was set up in 1988 by the Scandinavian Sleep Research Society. It consists of 21 questions on sleep, evaluating the past three months. The questions can be answered on a five-point scale, 1 to 5. It has been translated into Swedish and Danish.

Epworth Sleepiness Scale (ESS) ESS is a validated questionnaire assessing the probability of falling asleep in eight different situations in daily life with four alternative answers ranging from 0-3. The score ranges from 0-24, and the higher the score, the higher the level of daytime sleepiness. The ESS has been proven to correlate to the AHI in the Sleep Heart Health Study, showing higher levels of the ESS when the AHI was higher. There is also a correlation between the incidences of road traffic accidents and the ESS, as well as health-related questions relating to quality of life and the ESS. Daytime sleepiness is considered at a summary score of above 10. It has been translated into Swedish and Danish.

Short form 36 (SF-36) The SF-36 is a validated questionnaire that evaluates the quality of life in eight different health-related domains. It has been translated into Swedish and Danish.

Statistics A power calculation was performed based on Guimaraes et al.2009 results. The AHI was used in the calculation. Independent samples t-test, two-sided, anticipated effect size (Cohen's d) 0.8 (high), power ≥80%, probability level 5%. This gives a minimal sample size of 26 per group. The expected dropout of patients during the trial is 25% corresponding to a total of 9 patients in each group. To accommodate for this potential, the sample size was increased to 105 (35 in each group).

The study will use a prospective randomized open-blinded endpoint (PROBE) design with baseline measurements, intervention phase and follow-up measurements, and controls without intervention. Primary and secondary outcomes are values of AHI, snoring, BNSQ, ESS, and SF-36. These measures will be compared for baseline data and follow-up data by applying an independent-samples t-test, chi2 for proportion. ANCOVA will be used to estimate adjusted differences between the groups, adjusting for baseline values. Statistical analyses will be conducted using SPSS® version 28. A statistically significant level is defined as P<0,05.

Ethics The study has Ethical approval in Sweden and Denmark. The participants, men, and women, included in the study will be informed both orally and in written information before leaving informed consent. The participants can, without explanation, end the study without any negative impact on future care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with AHI 10 - 29 seeking for problems with snoring and obstructive sleep apnea, age 18 to 75.

Exclusion Criteria:

* Subjects with previous surgery of the soft palate, 9 < AHI > 29, smokers, New York Heart Association Functional Classification, NYHA ≥ 3. BMI >34,9.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 90 days. Between first measurement (inclusion in study at baseline) and second measurement (at follow-up after 90 days of intervention or serving as control)
  The primary outcome is the change in the apnea-hypopnea index (AHI) before and after three months of intervention or control.
  months of training with one of the modalities, according to two overnight ambulatory sleep apnea recordings.

SECONDARY OUTCOMES:
Questionnaires | 90 days. Between first measurement (inclusion in study at baseline) and second measurement (at follow-up after 90 days of intervention or serving as control)
  Change in results from questionnaires concerning snoring, the Basic Nordic Sleep Questionnaire (BNSQ). Daytime sleepiness assessed using the Epworth Sleepiness Scale (ESS) change in quality of life using the short form -36 (SF-36) after 3 months of training or control.
Snoring | 90 days. Between first measurement (inclusion in study at baseline) and second measurement (at follow-up after 90 days of intervention or serving as control)
  Change in snoring frequency and sound level dB (A) after 3 months of training or controls.
Tounge strength | 90 days. Between first measurement (inclusion in study at baseline) and second measurement (at follow-up after 90 days of intervention or serving as control)
  Change in muscle strength before and after treatment for 3 months of training or serving as controls. For measuring a device called IOPI, Iowa Oral Performance Instrument, is used.

CONTACTS AND LOCATIONS:
Overall Officials: Thorbjörn Holmlund, PhD, Principal Investigator — Region Västerbotten
Locations (3):
- Zealand University Hospital, Köge, Region Sjælland, Denmark
- Sweden (2):
  - Skåne University Hospital, Lund, Skåne County
  - Region Västerbotten, Umeå, Västerbotten County

IPD SHARING:
Plan to Share IPD: No
Data will be shared with other researchers upon request. The data will be anonymized before sharing to avoid being traced back to a single study participant.

REFERENCES:
- [Result] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Result] Franklin KA, Lindberg E. Obstructive sleep apnea is a common disorder in the population-a review on the epidemiology of sleep apnea. J Thorac Dis. 2015 Aug;7(8):1311-22. doi: 10.3978/j.issn.2072-1439.2015.06.11. PMID 26380759
- [Result] Wozniak DR, Lasserson TJ, Smith I. Educational, supportive and behavioural interventions to improve usage of continuous positive airway pressure machines in adults with obstructive sleep apnoea. Cochrane Database Syst Rev. 2014 Jan 8;(1):CD007736. doi: 10.1002/14651858.CD007736.pub2. PMID 24399660
- [Result] Lim J, Lasserson TJ, Fleetham J, Wright J. Oral appliances for obstructive sleep apnoea. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004435. doi: 10.1002/14651858.CD004435.pub3. PMID 16437488
- [Result] Svanborg E. Upper airway nerve lesions in obstructive sleep apnea. Am J Respir Crit Care Med. 2001 Jul 15;164(2):187-9. doi: 10.1164/ajrccm.164.2.2105010c. No abstract available. PMID 11463584
- [Result] Sunnergren O, Brostrom A, Svanborg E. Soft palate sensory neuropathy in the pathogenesis of obstructive sleep apnea. Laryngoscope. 2011 Feb;121(2):451-6. doi: 10.1002/lary.21371. PMID 21271605
- [Result] Jaghagen EL, Berggren D, Isberg A. Swallowing dysfunction related to snoring: a videoradiographic study. Acta Otolaryngol. 2000 Mar;120(3):438-43. doi: 10.1080/000164800750000702. PMID 10894423
- [Result] Levring Jaghagen E, Franklin KA, Isberg A. Snoring, sleep apnoea and swallowing dysfunction: a videoradiographic study. Dentomaxillofac Radiol. 2003 Sep;32(5):311-6. doi: 10.1259/dmfr/29209140. PMID 14709606
- [Result] Jaghagen EL, Berggren D, Dahlqvist A, Isberg A. Prediction and risk of dysphagia after uvulopalatopharyngoplasty and uvulopalatoplasty. Acta Otolaryngol. 2004 Dec;124(10):1197-203. doi: 10.1080/00016480410017954. PMID 15768818
- [Result] Jaghagen EL, Bodin I, Isberg A. Pharyngeal swallowing dysfunction following treatment for oral and pharyngeal cancer--association with diminished intraoral sensation and discrimination ability. Head Neck. 2008 Oct;30(10):1344-51. doi: 10.1002/hed.20881. PMID 18720519
- [Result] Camacho M, Certal V, Abdullatif J, Zaghi S, Ruoff CM, Capasso R, Kushida CA. Myofunctional Therapy to Treat Obstructive Sleep Apnea: A Systematic Review and Meta-analysis. Sleep. 2015 May 1;38(5):669-75. doi: 10.5665/sleep.4652. PMID 25348130
- [Result] Hagg M, Tibbling L. Effect of IQoro(R) training on impaired postural control and oropharyngeal motor function in patients with dysphagia after stroke. Acta Otolaryngol. 2016 Jul;136(7):742-8. doi: 10.3109/00016489.2016.1145797. Epub 2016 Feb 29. PMID 26924256
- [Result] Partinen M, Gislason T. Basic Nordic Sleep Questionnaire (BNSQ): a quantitated measure of subjective sleep complaints. J Sleep Res. 1995 Jun;4(S1):150-155. doi: 10.1111/j.1365-2869.1995.tb00205.x. PMID 10607192
- [Result] Arnardottir ES, Isleifsson B, Agustsson JS, Sigurdsson GA, Sigurgunnarsdottir MO, Sigurdarson GT, Saevarsson G, Sveinbjarnarson AT, Hoskuldsson S, Gislason T. How to measure snoring? A comparison of the microphone, cannula and piezoelectric sensor. J Sleep Res. 2016 Apr;25(2):158-68. doi: 10.1111/jsr.12356. Epub 2015 Nov 9. PMID 26553758
- [Result] Johns MW. Reliability and factor analysis of the Epworth Sleepiness Scale. Sleep. 1992 Aug;15(4):376-81. doi: 10.1093/sleep/15.4.376. PMID 1519015
- [Result] Sullivan M, Karlsson J, Ware JE Jr. The Swedish SF-36 Health Survey--I. Evaluation of data quality, scaling assumptions, reliability and construct validity across general populations in Sweden. Soc Sci Med. 1995 Nov;41(10):1349-58. doi: 10.1016/0277-9536(95)00125-q. PMID 8560302
- [Result] Baptista PM, Martinez Ruiz de Apodaca P, Carrasco M, Fernandez S, Wong PY, Zhang H, Hassaan A, Kotecha B. Daytime Neuromuscular Electrical Therapy of Tongue Muscles in Improving Snoring in Individuals with Primary Snoring and Mild Obstructive Sleep Apnea. J Clin Med. 2021 Apr 27;10(9):1883. doi: 10.3390/jcm10091883. PMID 33925376
- [Result] Al Ashry HS, Hilmisson H, Ni Y, Thomas RJ; APPLES Investigators. Automated Apnea-Hypopnea Index from Oximetry and Spectral Analysis of Cardiopulmonary Coupling. Ann Am Thorac Soc. 2021 May;18(5):876-883. doi: 10.1513/AnnalsATS.202005-510OC. PMID 33472017
- [Result] Zhang F, Tian Z, Shu Y, Zou B, Yao H, Li S, Li Q. Efficiency of oro-facial myofunctional therapy in treating obstructive sleep apnoea: A meta-analysis of observational studies. J Oral Rehabil. 2022 Jul;49(7):734-745. doi: 10.1111/joor.13325. Epub 2022 May 16. PMID 35342989
- [Result] Rueda JR, Mugueta-Aguinaga I, Vilaro J, Rueda-Etxebarria M. Myofunctional therapy (oropharyngeal exercises) for obstructive sleep apnoea. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD013449. doi: 10.1002/14651858.CD013449.pub2. PMID 33141943
- [Result] Torres-Castro R, Vilaro J, Marti JD, Garmendia O, Gimeno-Santos E, Romano-Andrioni B, Embid C, Montserrat JM. Effects of a Combined Community Exercise Program in Obstructive Sleep Apnea Syndrome: A Randomized Clinical Trial. J Clin Med. 2019 Mar 14;8(3):361. doi: 10.3390/jcm8030361. PMID 30875753